CLINICAL TRIAL: NCT02090478
Title: The Effect of Dietary Sugar Consumption on Sweet Taste Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Paul Wise, Associate Member, Monell Chemical Senses Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IND039A01WISE
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Sweet Taste Perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No change in dietary sugar levels (Sham Comparator): Group met with a dietician as often as the control group to discuss diet, but the dietician gave them advice geared toward no change in dietary sugar levels
  Interventions: Other: Sham diet manipulation
- Low sugar group (Experimental): Subjects met with a dietician who discussed diet records. After the first month (baseline, regular diet), the dietician made suggestions geared toward reducing calories from simple sugars by 40%. This will be achieved by replacing sugar calories with complex carbohydrates and fats, while maintaining energy balance (same number of calories as the baseline month).
  Interventions: Other: Low sugar diet

INTERVENTIONS:
Other: Low sugar diet — All subjects followed their usual diet during month 1. For months 2-4: sham diet intervention for the control group, 40% reduction in sugar calories for the experimental group. All subjects were allowed to chose any diet they wished during month 5.
  Arms: Low sugar group
Other: Sham diet manipulation — Subjects in the control group will meet with a dietician and discuss diet records, but the dietician will not instruct the control subjects to reduce the number of calories from simple sugars in the diet
  Arms: No change in dietary sugar levels

SUMMARY:
The purpose of the study is to determine how reducing the amount of simple sugars in the diet affects sweet taste perception. Healthy adult subjects will be assigned to either follow their usual diet, or to replace sugar calories with fats or starch.

The investigators hypothesize that eating less sugar will:

1. cause foods and drinks with a given amount of sugar to taste sweeter
2. cause people to prefer lower levels of sugar in foods and drinks

ELIGIBILITY:
Inclusion Criteria:

* Good general heath (by self report)
* Consume at least 2 sugar-containing soft drinks/day on average)
* Able to control diet (select their own foods)

Exclusion Criteria:

* Major illness of any kind within the last six months, or any chronic illness
* Daily use of medication, except for birth control, vitamins, and aspirin
* Regularly consume non-nutritive sweeteners
* Pregnant women
* Gained or lost 10% or more of their body weight in the last 3 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Sweet Taste Intensity over Five Months | Monthly (for five months)
  Subjects rated the sweetness of pudding and beverage samples that varied in sucrose concentration during each study month to determine how perception changes over time with diet manipulations
Change in Pleasantness Over Five Months | Monthly (five month participation duration total)
  Subjects rated hedonic value (degree to which the sample was pleasant) for model pudding and beverages that differed in concentration of sucrose once each month over five months to determine how perception changed over time with the diet manipulation

SECONDARY OUTCOMES:
Sucrose detection thresholds | Every month (for five months)
  Test of the minimum concentration of sucrose solution that subjects can discriminate from water. Forced-choice, ascending concentration method.
Body mass index | Every month (five months total)
  BMI, calculated based on weight and height. This was measured both to balance treatment groups and to ensure that assigned diets maintained adequate energy balance (no change in BMI over the study was the ideal outcome for all groups)
Diet records | Every month (five month total)
  Subject reported in detail the types and quantities of the foods and beverages they ate.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Wise, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Wise PM, Nattress L, Flammer LJ, Beauchamp GK. Reduced dietary intake of simple sugars alters perceived sweet taste intensity but not perceived pleasantness. Am J Clin Nutr. 2016 Jan;103(1):50-60. doi: 10.3945/ajcn.115.112300. Epub 2015 Nov 25. PMID 26607941